CLINICAL TRIAL: NCT02178176
Title: Participatory Design of Patient-centered Depression and Diabetes Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Hillary Bogner, Associate Professor, University of Pennsylvania
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1K18HS023445-01 (AHRQ)
Record Dates: First submitted 2014-06-26; First posted 2014-06-30 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Depression; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Depression; Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education, encouragement, card sort (Experimental)
  Interventions: Behavioral: Education, encouragement, card sort
- Education, encouragement (Active Comparator)
  Interventions: Behavioral: Education, encouragement

INTERVENTIONS:
Behavioral: Education, encouragement, card sort — Patients will identify factors involved in nonadherence. For each factor influencing adherence, the interventionist will engage the patient in a 4-step problem solving process.
  We will recognize patients' social and cultural context by addressing health-related priorities identified by the patient. The goal will be to identify those priorities which are likely to influence engagement in care and adherence to treatment. We will assess both biomedical (physical symptoms, diet and exercise) and nonbiomedical (financial, social and emotional) needs patients with Type 2 diabetes mellitus and depressive symptoms may wish to discuss in the context of their health. After the patients complete the card sort, interventionists will engage the patient in the 4-step problem solving process.
  Arms: Education, encouragement, card sort
Behavioral: Education, encouragement — Patients will identify factors involved in nonadherence. For each factor influencing adherence, the interventionist will engage the patient in a 4-step problem solving process.
  Arms: Education, encouragement

SUMMARY:
The burden of diabetes is anticipated to grow yet the proportion of adults whose diabetes is controlled is decreasing over time. This project can have a significant public health impact because we are refining and pilot testing a primary-care based intervention aimed at improving patient engagement and function which are critical components of diabetes care and are associated with improved glycemic control, lower disease-related health-care expenditures, and reduced mortality.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older
2. a current diagnosis of Type 2 DM
3. HbA1c 7%
4. current prescription for an oral hypoglycemic agent
5. able to communicate in English
6. willing to give informed consent

Exclusion Criteria:

1. acutely suicidal or psychotic (patients will not be randomized and PI or physician covering for PI will be paged immediately)
2. significant cognitive impairment at baseline (a total score on Mini-Mental State Examination (MMSE) 21)
3. markedly shortened life expectancy (diagnosis of metastatic cancer, end-stage renal disease on dialysis, or NYHA Class III or IV congestive heart failure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2013-09; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Depression: nine-item Patient Health Questionnaire (PHQ-9) | Baseline and 14 weeks
Glycemic control: hemoglobin A1c | Baseline and 14 weeks
Adherence to oral hypoglycemic agents: Medication Event Monitoring System | Over 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States